CLINICAL TRIAL: NCT01729351
Title: Comparative Effectiveness of Extrafine Hydrofluoroalkane Beclometasone Versus Fluticasone and Chlorofluorocarbon Beclometasone in Smoking Asthma - a Retrospective, Real-life Observational Study in a UK Primary Care Asthma Population
Brief Title: Qvar Therapy in Smoking Asthmatics
Status: Completed | Type: Observational
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Principal Investigator, David Price, Professor David Price, Research in Real-Life Ltd
Other Study IDs: R01911
Record Dates: First submitted 2012-11-09; First posted 2012-11-20 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Asthma; Smoking
Keywords: Primary Care; Particle size; beclomethasone dipropionate; Asthma Management; Maintenance Therapy; Metered-Dose Inhaler; Smoking
MeSH Terms: conditions — Asthma; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- IPDI EF HFA-BDP: Patients initiating inhaled corticosteroid therapy as extra-fine HFA-BDP MDI at the index date
- IPDI FP: Patients initiating inhaled corticosteroid therapy as FP via pMDI at the index date
- IPDI NEF HFA-BDP: Patients initiating inhaled corticosteroid therapy as non-extra-fine HFA-BDP via pMDI at the index date
- IPDA EF HFA-BDP: Patients increasing inhaled corticosteroid therapy as extra-fine HFA-BDP MDI at the index date
- IPDA FP: Patients increasing inhaled corticosteroid therapy as FP MDI at the index date
- IPDA NEF HFA-BDP: Patients initiating inhaled corticosteroid therapy as non-extra-fine HFA-BDP via pMDI at the index date

SUMMARY:
To evaluate the comparative effectiveness of extrafine hydrofluoroalkane beclometasone (EF HFA-BDP) and other inhaled corticosteroid (ICS) therapy commonly used in the UK, specifically fluticasone (FP) and non-extrafine (NEF) BDP (CFC-BDP and NEF HFA-BDP) in a UK primary care asthma population of current smokers.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-70 years
* Current smokers - explicitly coded in patient records or captured in patient questionnaires
* Evidence of asthma diagnosis and current therapy: ≥2 prescriptions for asthma at different points in time during the baseline year ± a diagnostic code for asthma
* On-going asthma therapy: ≥2 prescription for ICS during the outcome period (i.e. ≥1 prescription in addition to IPD prescription)
* ≥2 years continuous data (i.e. ≥1 year of baseline plus ≥1 year of outcome data)

Exclusion Criteria:

Patients will be excluded from the analysis if they have:

* Any chronic respiratory disease other than asthma
* Are prescribed:
* Maintenance oral steroid therapy during the baseline year
* Combination ICS/long-acting beta agonist (LABA) therapy during baseline year or at IPD
* Multiple ICS prescriptions at IPD or immediately before .

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are all current smokers ages between 16-70 years with evidence of asthma
Sampling Method: Non-Probability Sample
Enrollment: 7195 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Asthma Control proxy incorporating SABA use | 1 year
  Where control is defined as absence of:
  (i)Respiratory-related:
  Hospital attendance or admission A&E attendance, OR Out of hours attendance, OR Out-patient department attendance
  (ii)GP consultations for lower respiratory tract infection
  (iii)Prescriptions for acute courses of oral steroids
  (iv)Average prescribed daily dose of albuterol or terbutaline of ≤200mg
Asthma Exacerbations (ATS Definition) | 1 year
  Defined as an absence of the the following:
  1. Asthma related hospital attendance or admission, OR A&E attendance, OR
  2. Use of acute oral steroids.

SECONDARY OUTCOMES:
Exacerbation definition based on clinical experience | 1 year
  Defined as:
  (i)Respiratory-related:
  Hospital attendance / admissions OR A&E attendance OR Out of hours consultation OR GP consultation OR (ii) Use of acute oral steroids
Asthma control proxy excluding SABA usage | 1 year
  Control defined as absence of:
  (i) Respiratory-related:
  Hospital attendance or admission A&E attendance, OR Out of hours attendance, OR Out-patient department attendance
  (ii)GP consultations for lower respiratory tract infection
  (iii)Prescriptions for acute courses of oral steroids
Treatment Success | 1 year
  Success defined as:
  No respiratory-related:
  Hospital attendance or admission A&E attendance, OR Out of hours consultation, OR Out-patient department attendance
  No GP consultations for lower respiratory tract infection
  No prescriptions for acute courses of oral steroids
  No additional or change in therapy:
  Increased dose of ICS (≥50% increase), and/or Change in ICS and/or Change in delivery device, and/or Use of additional therapy as defined by: LABA, theophylline, leukotriene receptor antagonists (LTRAs).
Definite asthma-related hospitalisations | 1 year
  Hospitalisations coded with an asthma read code
ICS Compliance | 1 year
  Based on prescription refills
Incidence of oral thrust | 1 year
  Identified as:
  1. Topical oral anti-fungal prescriptions, and / or
  2. Coded for oral candidiasis
SABA Dose | 1 year
  Average daily dose of short-acting beta-agonist over the outcome year
Definite and probable asthma-related hospitalisations | 1 year
  Hospitalisations with an asthma read code + uncoded hospitalisations occurring within a 7-day window (either side of the hospitalisation date) of an asthma read code

CONTACTS AND LOCATIONS:
Overall Officials: David Professor Price, Principal Investigator — University of Aberdeen

REFERENCES:
- [Background] Price D, Martin RJ, Barnes N, Dorinsky P, Israel E, Roche N, Chisholm A, Hillyer EV, Kemp L, Lee AJ, von Ziegenweidt J, Colice G. Prescribing practices and asthma control with hydrofluoroalkane-beclomethasone and fluticasone: a real-world observational study. J Allergy Clin Immunol. 2010 Sep;126(3):511-8.e1-10. doi: 10.1016/j.jaci.2010.06.040. Epub 2010 Aug 9. PMID 20692026
- [Background] Barnes N, Price D, Colice G, Chisholm A, Dorinsky P, Hillyer EV, Burden A, Lee AJ, Martin RJ, Roche N, von Ziegenweidt J, Israel E. Asthma control with extrafine-particle hydrofluoroalkane-beclometasone vs. large-particle chlorofluorocarbon-beclometasone: a real-world observational study. Clin Exp Allergy. 2011 Nov;41(11):1521-32. doi: 10.1111/j.1365-2222.2011.03820.x. Epub 2011 Jul 14. PMID 21752116
- [Background] Hansell A, Hollowell J, Nichols T, McNiece R, Strachan D. Use of the General Practice Research Database (GPRD) for respiratory epidemiology: a comparison with the 4th Morbidity Survey in General Practice (MSGP4). Thorax. 1999 May;54(5):413-9. doi: 10.1136/thx.54.5.413. PMID 10212105
- [Background] Ivanova JI, Birnbaum HG, Hsieh M, Yu AP, Seal B, van der Molen T, Emani S, Rosiello RA, Colice GL. Adherence to inhaled corticosteroid use and local adverse events in persistent asthma. Am J Manag Care. 2008 Dec;14(12):801-9. PMID 19067497